CLINICAL TRIAL: NCT01046656
Title: Efficacy of Lactobacillus Reuteri DSM 17938 in the Prevention of Nosocomial Diarrhea in Children. Randomized Double-blind Placebo Controlled Trial
Brief Title: L Reuteri for the Prevention of Nosocomial Diarrhea
Acronym: PND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Hania Szajewska, Department of Paediatrics, The Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 152/2009; 152/2009
Record Dates: First submitted 2009-12-16; First posted 2010-01-12 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2009-12

CONDITIONS: Nosocomial Infection; Diarrhea; Gastroenteritis
Keywords: nosocomial infection; diarrhea; Lactobacillus reuteri; gastroenteritis; rotavirus
MeSH Terms: conditions — Cross Infection; Diarrhea; Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri (DSM 17938) — 5 drops once daily (10(8) CFU) for the entire duration of hospital stay

SUMMARY:
Nosocomial diarrhea is any diarrhea that a patient contracts in a health-care institution. In children, it is commonly caused by enteric pathogens, especially rotavirus. The reported incidence ranges from 4.5 to 22.6 episodes per 100 admissions. Nosocomial diarrhea may prolong the hospital stay and increase medical costs. One of the potential strategies for the prevention of nosocomial infections is the use of probiotics. The number of studies have shown the efficacy of Lactobacillus reuteri (DSM 17938) in the treatment of acute diarrhea. However, there are no data on the efficacy of L. reuteri in the prevention of nosocomial diarrhea. The investigators, therefore, plan to perform the study with the aim of evaluating the role of Lactobacillus reuteri DSM 17938 administration in the prevention of nosocomial gastroenteritis in a pediatric hospital setting.

DETAILED DESCRIPTION:
Infants will be randomly assigned at admission to receive L. reuteri in dose of 10(8) CFU in 5 drops of oil suspension or a comparable placebo once daily for the entire duration of their hospital stay.

Patients will be evaluated daily for stool number and consistency. In case of loose or watery stools occurring within 3 days after discharge, patients will be advised to contact hospital physicians. Stool samples obtained weekly and during an episode of diarrhea, will be analyzed for bacteria with standard stool cultures and rotavirus and adenovirus antigen.

ELIGIBILITY:
Inclusion Criteria:

* age 1-48 mo
* cause of hospitalization must be other than acute gastroenteritis or diarrhea

Exclusion Criteria:

* acute gastroenteritis within 3 days before admission
* other symptoms which suggest gastroenteritis
* usage of probiotics and/or prebiotics within 7 days before admission
* visible blood in the stool
* patient in bad condition
* lack of approval from patients parents
* breastfeeding
* no compliance

Ages: 1 Month to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Nosocomial diarrhea (passage of 3 or more loose or watery stools in a 24-hour period that will occur more than 72 hours after admission) | from 72nd hrs till the and of hospitalization no longer than 14 days

SECONDARY OUTCOMES:
Length of hospital stay in days | from 72nd hrs till the and of hospitalization no longer than 14 days
Recurrent diarrhea - recurrence of diarrhea after 48h of normal stools | from 72nd hrs till the and of hospitalization no longer than 14 days
Chronic diarrhea - diarrhea beyond 14 days | from 72nd hrs till the and of hospitalization no longer than 14 days
Diarrhea - the passage of 3 or more loose of watery stools in a 24 h period | from 72nd hrs till the and of hospitalization no longer than 14 days
Rotavirus infection - detection of rotavirus or antigen in the stools | from 72nd hrs till the and of hospitalization no longer than 14 days
Duration of diarrhea - time till the last loose watery stools from the onset of diarrhea measured in days) | from 72nd hrs till the and of hospitalization no longer than 14 days
Need for rehydration | from 72nd hrs till the and of hospitalization no longer than 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical University of Warsaw, Department of Paediatrics, Warsaw, Poland

REFERENCES:
- [Derived] Wanke M, Szajewska H. Lack of an effect of Lactobacillus reuteri DSM 17938 in preventing nosocomial diarrhea in children: a randomized, double-blind, placebo-controlled trial. J Pediatr. 2012 Jul;161(1):40-3.e1. doi: 10.1016/j.jpeds.2011.12.049. Epub 2012 Feb 4. PMID 22306046